CLINICAL TRIAL: NCT00888615
Title: A Phase II Evaluation of Elesclomol Sodium and Weekly Paclitaxel in the Treatment of Recurrent or Persistent Platinum-Resistant Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Elesclomol Sodium and Paclitaxel in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0260; NCI-2011-01919 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000641202; GOG-0260; GOG-0260 (Other: NRG Oncology); GOG-0260 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Tumor; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — elesclomol; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel, elesclomol sodium) (Experimental): Patients receive paclitaxel IV over 1 hour and elesclomol sodium IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. NOTE: Patients who are currently on treatment must not be dosed with elesclomol sodium after 12/31/2015. All other study procedures, with the exception of elesclomol sodium administration and paclitaxel administration, should continue in accordance with protocol requirements. Any treatment given after 12/31/2015, including continuation of paclitaxel, will be considered off study.
  Interventions: Drug: Elesclomol Sodium; Drug: Paclitaxel

INTERVENTIONS:
Drug: Elesclomol Sodium — Given IV
  Other Names: STA-4783
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase II trial studies how well elesclomol sodium and paclitaxel work in treating patients with ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer that has returned after a period of improvement (recurrent) or is persistent. Drugs used in chemotherapy, such as elesclomol sodium and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Elesclomol sodium may also help paclitaxel work better by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the antitumor activity of elesclomol (elesclomol sodium) and paclitaxel in patients with persistent or recurrent ovarian, fallopian tube, or primary peritoneal cancer primarily through the frequency of objective tumor responses.

II. To determine the nature and degree of toxicity of elesclomol and paclitaxel in this cohort of patients.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival and overall survival of patients treated with elesclomol and paclitaxel.

OUTLINE:

Patients receive paclitaxel intravenously (IV) over 1 hour and elesclomol sodium IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: Patients who are currently on treatment must not be dosed with elesclomol sodium after 12/31/2015. All other study procedures, with the exception of elesclomol sodium administration and paclitaxel administration, should continue in accordance with protocol requirements. Any treatment given after 12/31/2015, including continuation of paclitaxel, will be considered off study.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report

  * Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's tumor, or adenocarcinoma not otherwise specified (N.O.S.)
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III protocol for the same patient population
* Patients must have a GOG performance status of 0, 1, or 2
* Patients must have baseline lactate dehydrogenase (LDH) levels =< 0.8 x upper limit of normal (ULN)
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy directed at the malignant tumor, including biological and immunologic agents, must be discontinued at least three weeks prior to registration
* Prior therapy

  * Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment
  * Patients must have NOT received any additional cytotoxic chemotherapy for management of recurrent or persistent disease, including retreatment with initial chemotherapy regimens; (Note: optimal evaluation of the safety and efficacy of new chemotherapy regimens is best performed in patients with minimal prior therapy; non-investigational therapy, such as retreatment with platinum and/or paclitaxel, is non-curative in the setting of recurrent disease, and can generally be safely administered to patients following participation in a phase II trial)
  * Patients are allowed to receive, but are not required to receive, one additional non-cytotoxic regimen for management of recurrent or persistent disease according to the following definition:
  * Non-cytotoxic (biologic or cytostatic) agents include (but are not limited to) hormones, monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction
  * Patients must be considered platinum resistant or refractory according to standard GOG criteria, i.e., have had a treatment-free interval following platinum of less than 6 months, or have progressed during platinum-based therapy
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Neurologic function: neuropathy (sensory and motor) less than or equal to Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test prior to study entry and be practicing an effective form of contraception
* Cautions and prohibited medications/treatments

  * Since elesclomol is a substrate for cytochrome P450 family 2, subfamily C, polypeptide 9 (CYP2C9), cytochrome P450 family 2, subfamily D, polypeptide 6 (CYP2D6), cytochrome P450 family 2, subfamily C, polypeptide 19 (CYP2C19), and cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) and an inducer of CYP3A4, cytochrome P450 family 1, subfamily A, polypeptide 2 (CYP1A2), cytochrome P450 family 2, subfamily A, polypeptide 6 (CYP2A6), and cytochrome P450 family 2, subfamily E, polypeptide 1 (CY2E1), it is recommended that the following be used with caution: sensitive substrates of CYP3A4, CYP1A2, and CY2E1, and strong inhibitors and inducers of CYP2C9, CYP2D6, CYP2C19, and CYP3A4

Exclusion Criteria:

* Patients who have had prior therapy with elesclomol or prior second-line cytotoxic chemotherapy
* Patients who have received radiation to more than 25% of marrow-bearing areas
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Monk, Principal Investigator — NRG Oncology
Locations (163):
- United States (163):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California San Diego, San Diego, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Piedmont Hospital, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Stony Brook University Medical Center, Stony Brook, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - University of Toledo, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin

REFERENCES:
- [Derived] Monk BJ, Kauderer JT, Moxley KM, Bonebrake AJ, Dewdney SB, Secord AA, Ueland FR, Johnston CM, Aghajanian C. A phase II evaluation of elesclomol sodium and weekly paclitaxel in the treatment of recurrent or persistent platinum-resistant ovarian, fallopian tube or primary peritoneal cancer: An NRG oncology/gynecologic oncology group study. Gynecol Oncol. 2018 Dec;151(3):422-427. doi: 10.1016/j.ygyno.2018.10.001. Epub 2018 Oct 8. PMID 30309721

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
Started | 58
Completed | 56
Not Completed | 2
Not completed — No treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
Number analyzed (Participants) | 56
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0
  30-39 years | 0
  40-49 years | 6
  50-59 years | 12
  60-69 years | 22
  70-79 years | 14
  >= 80 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 0
Cell Type [Count of Participants; unit: Participants]
  Adenocarcinoma, nos | 8
  Clear cell | 2
  Endometrioid | 2
  Serous | 44

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Objective Response
Description: Proportion of Participants with Object Response (per response evaluation criteria in solid tumors criteria (RECIST V1.1) for target lesions as assessed by MRI: Complete Response (CR), disappearance of all target lesions, Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
Number analyzed (Participants) | 56
Proportion of participants | 0.196 [0.114 to 0.304]

2. Primary Outcome: Duration of Objective Response
Description: Duration of objective response (months)
Time Frame: Up to 5 years
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
Number analyzed (Participants) | 56
months | 9.2 [5.5 to 14.9]

3. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: The frequency of patients who experienced at least one adverse effect (with a grade of 1 or higher). Adverse effects are defined as any unfavorable and unintended sign, symptom, or disease that occurs in a patient administered a medical treatment, whether the event is considered related or unrelated to the medical treatment.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
Number analyzed (Participants) | 56
Participants | 56

4. Primary Outcome: The Number of Participants Who Experienced at Least One Grade 3 Adverse Event
Description: The number of participants who experienced at least one grade three (or higher) adverse effect. The severity of observed adverse effects is graded using the NCI CTCAE version 4.0.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
Number analyzed (Participants) | 56
Participants | 26

5. Secondary Outcome: Progression-free Survival (Median)
Description: Progression-free survival (median, in months) will be analyzed by Kaplan-Meier analysis (progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions (also a 5 mm absolute increase is also required), or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
Number analyzed (Participants) | 56
months | 3.6 [2.03 to 5.65]

6. Secondary Outcome: Overall Survival (Median)
Description: Overall survival (median, in months) will be analyzed by Kaplan-Meier analysis.
Time Frame: From start of treatment to time of death or the date of last contact, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
Number analyzed (Participants) | 56
months | 13.3 [10.38 to 19.45]

ADVERSE EVENTS:
Arm/Group | Treatment (Paclitaxel, Elesclomol Sodium)
All-Cause Mortality (participants affected / at risk) | 43/56
Serious Adverse Events (participants affected / at risk) | 18/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Elesclomol Sodium) (N=56)
Atrial Fibrillation (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Colonic Hemorrhage (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Skin Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Elesclomol Sodium) (N=56)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 53
Supraventricular Tachycardia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Cardiac Disorders - Other (Cardiac disorders) | 1
Ventricular Arrhythmia (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 2
Chest Pain - Cardiac (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Hearing Impaired (Ear and labyrinth disorders) | 2
Watering Eyes (Eye disorders) | 1
Flashing Lights (Eye disorders) | 1
Blurred Vision (Eye disorders) | 3
Floaters (Eye disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 2
Colonic Obstruction (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 25
Diarrhea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 15
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 7
Stomach Pain (Gastrointestinal disorders) | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 22
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Oral Dysesthesia (Gastrointestinal disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 6
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 30
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 2
Pain (General disorders) | 5
Flu Like Symptoms (General disorders) | 1
Edema Limbs (General disorders) | 9
Facial Pain (General disorders) | 1
Edema Face (General disorders) | 1
Fatigue (General disorders) | 41
Fever (General disorders) | 8
Gait Disturbance (General disorders) | 1
Chills (General disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 4
Tooth Infection (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 2
Nail Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Esophageal Infection (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 8
Bronchial Infection (Infections and infestations) | 3
Enterocolitis Infectious (Infections and infestations) | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Investigations - Other (Investigations) | 2
Weight Loss (Investigations) | 3
Weight Gain (Investigations) | 4
Platelet Count Decreased (Investigations) | 10
Lymphocyte Count Decreased (Investigations) | 5
Ejection Fraction Decreased (Investigations) | 1
Creatinine Increased (Investigations) | 7
Cholesterol High (Investigations) | 3
Neutrophil Count Decreased (Investigations) | 27
Blood Bilirubin Increased (Investigations) | 2
White Blood Cell Decreased (Investigations) | 37
Aspartate Aminotransferase Increased (Investigations) | 5
Alkaline Phosphatase Increased (Investigations) | 9
Alanine Aminotransferase Increased (Investigations) | 8
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 14
Hypokalemia (Metabolism and nutrition disorders) | 11
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 18
Hypercalcemia (Metabolism and nutrition disorders) | 1
Glucose Intolerance (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 22
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tremor (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 30
Peripheral Motor Neuropathy (Nervous system disorders) | 4
Paresthesia (Nervous system disorders) | 4
Neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Extrapyramidal Disorder (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 2
Concentration Impairment (Nervous system disorders) | 1
Akathisia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 14
Depression (Psychiatric disorders) | 9
Delirium (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 5
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 1
Urinary Urgency (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 3
Urinary Frequency (Renal and urinary disorders) | 6
Proteinuria (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Chronic Kidney Disease (Renal and urinary disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Laryngopharyngeal Dysesthesia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Scalp Pain (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3
Nail Ridging (Skin and subcutaneous tissue disorders) | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 3
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 25
Thromboembolic Event (Vascular disorders) | 3
Lymphedema (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Hot Flashes (Vascular disorders) | 5
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less